CLINICAL TRIAL: NCT04849611
Title: Covid-19 Fear and Compliance With Protective Measures of Students Continuing Face-to-Face Education in the Covid-19 Pandemic Process
Brief Title: Covid-19 Fear and Compliance With Protective Measures of Students
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hacer Gok Ugur, Public Health Nursing Department, Ordu University
Other Study IDs: q9wrjg2p
Record Dates: First submitted 2021-03-22; First posted 2021-04-19 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Covid-19
Keywords: Covid-19; School; Student; Fear; Protective Measure
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was carried out to determine the fear of Covid-19 and the compliance with protective measures of students who continue their education face-to-face during the covid-19 pandemic process.

DETAILED DESCRIPTION:
The study was carried out descriptively. The study population of a province pandemic period junior ongoing training to face in Turkey. Sample constituted reached 188 students with snowball sampling method. The data of the study were collected using the "Questionnaire Form" prepared by the researchers and the "Covid-19 Fear Scale". Data collection tools were applied to the participants electronically via Google Forms.

ELIGIBILITY:
Inclusion Criteria:

Students who volunteered to participate in the study, had their parents' consent, had a web-based smart device, and continued face-to-face education were included.

Exclusion Criteria:

-

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: continued face-to-face education students
Sampling Method: Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Covid-19 Fear | November-March
  Covid-19 Fear Scale: The scale developed by Ahorsu et al. (2020) was adapted to Turkish by Bakioglu, Korkmaz and Ercan (2020). The scale, consisting of seven questions, is a 5-point Likert (1: Strongly disagree, 5: Strongly agree) type. The scale consists of one dimension. The scores that can be obtained from the scale range from 7 to 35. The total score obtained from all items of the scale reflects the level of Covid-19 fear experienced by the individual. A high score means experiencing a high level of fear.

OTHER OUTCOMES:
Information Form | November-March
  The form consists of two parts. In the first part, there are 14 questions that determine the socio-demographic characteristics of the students (age, gender, class, family type, mother education, father education, monthly income level, knowledge about Covid-19, information source, catching Covid-19, family's catching Covid-19, worrying about the family in terms of the illness, thinking that they can be protected from Covid-19 and being knowledgeable about the methods of protection from Covid-19). In the second part, the practices of students on protection methods from Covid-19 were prepared within the framework of mask (14 questions), hand washing (8 questions) and social distance (17 questions) measures. No scoring will be made in this section. Students' compliance with protective measures will be evaluated as "yes" "no" "sometimes".

CONTACTS AND LOCATIONS:
Overall Officials: Hacer GOK UGUR, Assoc. Prof., Principal Investigator — Ordu University
Locations (1):
- Ordu University, Ordu, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahorsu DK, Lin CY, Imani V, Saffari M, Griffiths MD, Pakpour AH. The Fear of COVID-19 Scale: Development and Initial Validation. Int J Ment Health Addict. 2022;20(3):1537-1545. doi: 10.1007/s11469-020-00270-8. Epub 2020 Mar 27. PMID 32226353
- [Background] Bakioglu F, Korkmaz O, Ercan H. Fear of COVID-19 and Positivity: Mediating Role of Intolerance of Uncertainty, Depression, Anxiety, and Stress. Int J Ment Health Addict. 2021;19(6):2369-2382. doi: 10.1007/s11469-020-00331-y. Epub 2020 May 28. PMID 32837421